CLINICAL TRIAL: NCT00005741
Title: Indigenous Outreach Among Injection Drug Users to Treat and Control TB
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4950; R01HL055760 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-05

CONDITIONS: Lung Diseases; Tuberculosis
MeSH Terms: conditions — Lung Diseases; Tuberculosis

SUMMARY:
The Community Outreach Intervention Project (COIP) implemented and evaluated a TB intervention with injection drug users (IDUs) in two Chicago Neighborhoods, guided by the indigenous outreach leadership model that had been used for AIDS prevention among drug users.

DETAILED DESCRIPTION:
BACKGROUND:

Tuberculosis was on the decline from the mid 1950s until the mid 1980s; however, the United States is now experiencing a resurgence of tuberculosis. In 1992, approximately 27,000 new cases were reported, an increase of about 20 percent from 1985 to 1992. Not only are tuberculosis cases on the increase, but a serious aspect of the problem is the recent occurence of outbreaks of multidrug resistant (MDR) tuberculosis, which poses an urgent public health problem and requires rapid intervention.

Control programs involve two major components. First, and of highest priority, is to detect persons with active tuberculosis and treat them with effective antituberculosis drugs, which prevents death from tuberculosis and stops the transmission of infection to other persons. Treatment of active tuberculosis involves taking multiple antituberculosis drugs daily or several times weekly for at least six months. Failure to take the medications for the full treatment period may mean that the disease is not cured and may recur. If sufficient medications are not prescribed early and taken regularly, the tuberculosis organism can become resistant to the drugs, and the drug resistant tubercuosis then may be transmitted to other persons. Drug resistant disease is difficult and expensive to treat, and in some cases, cannot be treated with available medications.

The second major goal of control efforts is the detection and treatment of persons who do not have active tuberculosis, but who have latent tuberculosis infection. These people may be at high risk of developing active tuberculosis. The only approved treatment modality for preventive therapy requires treatment daily or twice weekly for a minimum of six months, and many patients do not complete the full course of therapy. Public and patient programs are needed to increase the awareness of the problems associated with tuberculosis control.

The study is part of the NHLBI initiative "Behavioral Interventions for Control of Tuberculosis" . The concept for the initiative originated from the National Institutes of Health Working Group on Health and Behavior. The Request for Applications was released in October, 1994.

DESIGN NARRATIVE:

Three hypotheses were tested. The first was that rates of treatment adherence would be greater among actively infected injection drug users assisted through indigenous outreach than through conventional TB control methods practiced by the Chicago Department of Health. The second hypothesis was that rates of compliance with contact tracing, screening and treatment wouldl be greater through the COIP intervention than through the practices of the Health Department. The third was that community level rates of TB would decrease over the years of the study as a result of the intervention.

Enrollment of the cases and contacts for Phase II began in July 1996. The intervention was implemented by a specially trained indigenous outreach staff guided by an experienced ethnographer. Quantitative and qualitative methods were used to assess the effects of the intervention on treatment completion, attendance, compliance with contact and screening efforts, knowledge of TB transmission, reduction of health risk behavior and rates of TB infection.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2001-08 (Actual)